CLINICAL TRIAL: NCT05577442
Title: Peking University Cancer Hospital & Institute
Brief Title: Trastuzumab, Pyrotinib Combined With Dalpiciclib and Endocrine Therapy for HR +/HER2 + Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Li Huiping, Head of the department of breast oncology, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BC-Ⅱ-077
Record Dates: First submitted 2022-10-09; First posted 2022-10-13 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Breast Neoplasm Female
MeSH Terms: interventions — Trastuzumab; dalpiciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trastuzumab, Pyrotinib Combined With Dalpiciclib and Endocrine Therapy (Experimental): for the HR+/HER2+MBC will be treated with Trastuzumab, Pyrotinib Combined With Dalpiciclib and Endocrine Therapy. Endocrine drug be determined by physician depend on the history.
  Interventions: Drug: Trastuzumab, Pyrotinib Combined With Dalpiciclib and Endocrine Therapy

INTERVENTIONS:
Drug: Trastuzumab, Pyrotinib Combined With Dalpiciclib and Endocrine Therapy — Trastuzumab (8-6mg/3weekly)，Pyrotinib（320mg/day）Dalpiciclib（125mg/day，With three weeks separated by one week）
  Other Names: Trastuzumab Pyrotinib Dalpiciclib

SUMMARY:
This study investigates the efficacy and safety of trastuzumab, pyrotinib combined with dalpiciclib and endocrine therapy for patients with advanced HR+/HER2+ brest cancer, providing more possible effective regimens for the survival benefit of these patients in clinical practice.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, multicenter, phase II clinical study. Subjects were eligible for screening and entered the trial period after enrollment and received treatment with pyrotinib（320mg/day), trastuzumab(8 mg→6mg/every 3 week), dalpiciclib(125mg once daily for 3 weeks, followed by 1 week off in each 4-week cycle), endocrine therapy until disease progression, or intolerable toxicity, or withdrawal of informed consent, or discontinuation of medication at the investigator 's discretion. On-study imaging assessments were performed according to RECIST 1.1 criteria and the site assessment was final.

ELIGIBILITY:
Inclusion Criteria:

1. Female breast cancer patients of any menopausal status aged 18-75 years.
2. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
3. Female breast cancer patients with HER2-positive HR-positive of recurrence or metastasis and are not suitable for surgical resection or radiation therapy with the purpose of cure.
4. ER and/or PR +: defined as positively stained tumor cells representing ≥ 10% of all tumor cells (confirmed by investigator review at the site) and HER2 +: defined as IHC 3 + or IHC 2 + and FISH +/CISH +.
5. measurable lesions by RECIST 1.1 criteria.
6. Patients' previous treatment should meet: a) prior systemic (neo) adjuvant therapy is allowed but not required, and if received, the disease-free interval (DFI) must be > 24 months (DFI is defined as the time from surgery to the first recurrence); b) ≤ 1 line of systemic therapy for the tumor (including anti-HER2 targeted therapy, endocrine therapy and chemotherapy) is received at the metastatic stage;
7. Stable patients with brain metastases are allowed.
8. life expectancy ≥ 12 weeks.
9. adequate organ and bone marrow function.
10. adequate cardiac reserve, left ventricular ejection fraction (LVEF) ≥ 45% on echocardiogram.

Exclusion Criteria:

1. patients who are not suitable for endocrine therapy as judged by the investigator. Including symptomatic, advanced patients with disseminated visceral disease who are at short-term risk of life-threatening complications (including patients with uncontrolled large exudates [pleural, pericardial, abdominal], pulmonary lymphangitis and more than 50% hepatic involvement).
2. previous treatment with CDK4/6 inhibitors.
3. previous treatment with TKI.
4. visceral crisis.
5. Major surgery, chemotherapy, radiation therapy, any investigational agent, or other anticancer therapy within 2 weeks before entering the study.
6. Have been diagnosed with any other malignancy within 3 years before entering the study, except for curatively treated non-melanoma skin cancer, basal cell or squamous cell skin cancer, or cervical carcinoma in situ.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-10-20 (Estimated); Primary Completion 2023-10-20 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
ORR | 8week

IPD SHARING:
Plan to Share IPD: Undecided